CLINICAL TRIAL: NCT02396433
Title: Phase I/II Clinical Trial of the Combination of Carboplatin, Eribulin Mesylate, and E7449 in Patients With BRCA-Related Cancers
Brief Title: Combination of Carboplatin, Eribulin Mesylate, and E7449 in BRCA-Related Cancers
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: lack of funding.
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, Virginia G. Kaklamani, Professor of Medicine Hematology/ Oncology, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTMS# 14-2024
Record Dates: First submitted 2015-02-10; First posted 2015-03-24 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Cancer of the Breast
Keywords: Halaven; BRCA; E7449
MeSH Terms: conditions — Breast Neoplasms | interventions — Carboplatin; eribulin; stenoparib; Poly(ADP-ribose) Polymerase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carboplatin, eribulin, and E7449 (Experimental): This is a phase I/II clinical trial of the combination of carboplatin, eribulin, and E7449.
  Interventions: Drug: Carboplatin; Drug: Eribulin; Drug: E7449

INTERVENTIONS:
Drug: Carboplatin — Carboplatin will be given on day 1 of each cycle.
  Other Names: Paraplatin
Drug: Eribulin — Eribulin will be given on days 1 and 8 of each cycle.
  Other Names: Halaven
Drug: E7449 — E7449 will be given daily (days 1-21) during each cycle. Patients will continue to receive treatment until progression of disease or discontinuation due to unacceptable side effects.
  Other Names: PARP inhibitor

SUMMARY:
Non-randomized, open-label, multi-center, phase I/II, dose-escalation study of the combination of carboplatin, eribulin, and E7449.

DETAILED DESCRIPTION:
This is a phase I/II clinical trial of the combination of carboplatin, eribulin, and E7449. A cycle will be defined as 21 days. Carboplatin will be given on day 1 of each cycle. Eribulin will be given on days 1 and 8 of each cycle. E7449 will be given daily (days 1-21) during each cycle. Patients will continue to receive treatment until progression of disease or discontinuation due to unacceptable side effects.

ELIGIBILITY:
Inclusion Criteria:

Phase I only

* Patients must have stage IV breast or ovarian cancer or another BRCA mutation-related cancer.
* Patients may have either measurable or evaluable disease per RECIST 1.1 criteria.

NOTE: Measurable lesions are defined as those that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan.

* Patients must be refractory to / intolerant of established therapy known to provide clinical benefit for their condition.

Both Phase I & II

* Patients must have archival biopsy specimens (preferably from metastatic disease) available for research tests. If a suitable biopsy specimen is not available, patients will be asked to undergo a research biopsy to procure tissue.
* Patients must be ≥ 18 years.
* Females of childbearing potential must not have had unprotected sexual intercourse within 30 days prior to study entry and must agree to use a highly effective method of contraception. Females who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 4 weeks prior to dosing and must continue to use the same contraceptive during the study and for 30 days after study drug discontinuation
* Patients must have an ECOG performance status 0-1.
* Patients may have had a prior diagnosis of cancer if it has been > 5 years since their last treatment for that cancer.
* Patients must have normal organ and marrow function as defined below:

Leukocytes ≥ 3,000/μL Absolute neutrophil count ≥ 1,500/μL Platelets ≥ 100,000/μL Creatinine within normal limits or creatinine clearance ≥30

* Patients must be able to swallow and retain oral medication.
* Patients who were receiving prior systemic therapy: Prior treatment related side effects must have resolved to < Grade 2 severity (except alopecia and infertility).
* All patients must have given signed, informed consent prior to registration on study.

Phase II Only

* Patients must have stage IV breast or ovarian cancer
* Patients must have BRCA1/2 deleterious mutations, PTEN deficiency, or cancer with a high HRD score as assessed by Myriad's assay
* Patients must have measurable disease per RECIST 1.1 criteria (see above for definition).
* Patients may not have received more than 3 chemotherapeutic regimens for metastatic disease.
* Patients who may not have received treatment with prior carboplatin, eribulin or a PARP inhibitor.

Exclusion Criteria:

* Women who are pregnant or lactating are not eligible
* Patients who are undergoing concomitant radiotherapy are not eligible.
* Patients who are receiving any other investigational agents or concurrent anticancer therapy are not eligible.

NOTE: Previous systemic treatment is allowed with a 14 day (Phase I) or 21 day (Phase II) washout period prior to registration.

* Patients who are taking any herbal (alternative) medicines are not eligible. Patients must be off any such medications by the time of registration.
* Patients with known brain metastases are not eligible for participation unless the following are met:

Brain metastases are treated (either with surgical excision, stereotactic radiosurgery or radiotherapy and have been stable for at least 4 weeks (MRI documented) Patient is asymptomatic and has discontinued corticosteroids if taken for that purpose

Patients with any of the following conditions or complications are NOT eligible for participation:

GI tract disease resulting in an inability to take oral medication Malabsorption syndrome Require IV alimentation History of prior surgical procedures affecting absorption Uncontrolled inflammatory GI disease (e.g., Crohn's, ulcerative colitis). Hypersensitivity of any of the components of E7449, carboplatin, eribulin History of significant neurological (no neuropathy > Grade 2) or psychiatric disorders.

Significant non-neoplastic liver disease (e.g., cirrhosis, active chronic hepatitis).

Significant non-neoplastic renal disease. Immunocompromised subjects, including subjects known to be infected with human immunodeficiency virus (HIV).

Uncontrolled endocrine diseases (e.g., diabetes mellitus, hypothyroidism or hyperthyroidism, adrenal disorder) i.e., requiring relevant changes in medication within the last month or hospital admission within the last three months Active infection requiring systemic therapy. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, uncontrolled arterial hypertension, unstable angina, myocardial infarction or stroke within 6 months of the first dose of study drug; or cardiac arrhythmia requiring medical treatment.

Prolongation of QTc interval to > 480 msec when electrolytes balance is normal. Major surgery within 4 weeks prior to the first dose of study drug

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Safety of E7449 will be measured by the number, frequency and severity of adverse events. | Baseline to 24 months
  Patients will be evaluated by MD at clinic visits during Cycle 1, on Day 1 of all 21-day cycles, and will have additional evaluations if clinically indicated.
MTD (maximum tolerated dose) of E7449 will be measured by the number, frequency and severity of adverse events. | Baseline to 21 days
  Maximum tolerated dose (MTD) defined as highest dose studied in which the incidence of non-hematologic DLT (dose limiting toxicity) is defined as any Grade ≥ 3 toxicity, and a hematologic DLT is defined as any Grade ≥ 4 toxicity, both by CTCAE v 4.03 criteria.

SECONDARY OUTCOMES:
Overall response rate will be measured by the evaluation of target and non-target lesions for changes in tumor measurements. | Baseline to first occurrence of disease progression or death. (up to 6 weeks)
  The overall response rate (ORR) will be defined as response after scans (CT or MRI) assessed after two cycles of therapy (1 cycle = 3 weeks).

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Kaklamani, Principal Investigator — UTHSCSA@CTRC